CLINICAL TRIAL: NCT06010238
Title: Short Term Variation Analysis Versus Visual Evaluation of Cardiotocography in Fetal Growth Restriction
Brief Title: STV Analysis Versus Visual Evaluation of Cardiotocography in FGR
Acronym: SAVEFGR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Wessel Ganzevoort, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 84591
Record Dates: First submitted 2023-07-21; First posted 2023-08-24 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Fetal Growth Retardation
Keywords: fetal growth restriction; cardiotocography; perinatal death; short term variation
MeSH Terms: conditions — Fetal Growth Retardation; Perinatal Death

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual interpretation of cardiotocography (Active Comparator): Monitoring by visual interpretation of cardiotocography
  Interventions: Device: Visual interpretation
- Short term variation (Experimental): Short term variation by computer software analysis
  Interventions: Device: Short term variation

INTERVENTIONS:
Device: Short term variation — Short term variation in computer software analysis
  Arms: Short term variation
Device: Visual interpretation — Visual interpretation of cardiotocography
  Arms: Visual interpretation of cardiotocography

SUMMARY:
This stepped wedge cluster randomized clinical trial investigates whether in pregnant women with severe, early-onset fetal growth restriction, the use of STV analysis in fetal monitoring improves the chances of perinatal survival, compared with visual evaluation of the cardiotocography.

DETAILED DESCRIPTION:
Severe, early-onset fetal growth restriction (FGR, <32 weeks gestation) is a condition in which the fetus does not reach its growth potential due to placental insufficiency[. This condition affects about 0.3% of pregnancies, accounting for an estimated 15,000 babies in Europe being born premature below 32 weeks gestation. The main clinical dilemma of FGR lies in the timing of birth, given the balance of risks of antenatal mortality and severe damage to organs and the aggravated neonatal effects of prematurity: death or survival with severe neurodevelopmental impairment. The mainstay of clinical management in these cases pivots around the anticipation of the risk of fetal demise from placental oxygenation failure. The monitoring variables that are currently available comprise assessment of the severity of metabolic insufficiency (fetal size and growth, Doppler ultrasound, serum biomarkers) and the early detection of progressive fetal hypoxia with cardiotocography (CTG). The common approach is to deliver the fetus when signs of advanced hypoxia appear on CTG. A delicate balance exists between having the fetus born (too) early and facing the risks of extreme prematurity combined with a very low birthweight; and between delivering the fetus (too) late when the fetus has the disadvantage of hypoxia at birth. The decision when to deliver the fetus, is made mostly based on the CTG. The inter- and intra-observer variability could be overcome by software analysis according to the original Dawes&Redman algorithm. The software calculates the short-term variation (STV) of the inter-beat interval expressed in milliseconds, and a range of secondary calculations. In contrast with repeated decelerations, when fetal hypoxia is considered evident, the place of the software analysis of the fetal heart rate variability is less clear. Although the advantages of mathematized and uniform quantification of the fetal heart rate variability appear self-evident, there are no studies with sufficient power to detect an association of intervention based on STV at any threshold with the most important outcomes: fetal death and long-term infant outcome.

The purpose of this study is to assess the outcomes of monitoring the fetal condition with STV in computerized CTG compared to visual interpretation of the CTG in order to time delivery in pregnant women with severe, early-onset FGR.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a singleton pregnancy between 24 weeks and 0 days and 31 weeks and 6 days with severe, early-onset fetal growth restriction, admitted in hospital or frequently evaluated ambulatory by CTG (according to local protocol) for fetal monitoring.
* Fetal growth restriction is defined in line with the international Delphi consensus as biometric ultrasound measurement of the abdominal circumference (AC) OR a combination of measurements resulting in an estimated fetal weight (EFW) below the 3rd percentile (<p3) OR a combination of EFW <p10 AND uterine artery pulsatility index (PI) >p95 OR umbilical artery Doppler PI >p95.
* Maternal age ≥ 18 years.
* Able to provide written informed consent for collection and use of data on informed consent form in available language.

Exclusion Criteria:

* Known congenital or chromosomal anomalies influencing perinatal outcome.
* Imminent labour or expected maternal indication for delivery < 48 hours.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 800 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of pregnancies resulting in perinatal death | Before discharge from neonatal intensive care unit (NICU), up to 1 year
  Perinatal death is defined as antenatal death or neonatal/infant death before discharge from NICU

SECONDARY OUTCOMES:
Proportion of children with major neonatal morbidity | Before discharge from NICU, up to 1 year
  Major neonatal morbidity is a composite outcome defined as intraventricular hemorrhage grade 3 or more, periventricular leukomalacia grade 2 or more, moderate or severe bronchopulmonary dysplasia, necrotizing enterocolitis Bell stage 2 or more, or retinopathy of prematurity requiring therapy.
Proportion of children with neonatal morbidities | Before discharge from NICU, up to 1 year
  Individual neonatal morbidities of the abovementioned composite outcome and additionally persisting ductus arteriosus, persistent pulmonary hypertension of the newborn (PPHN), respiratory distress syndrome (RDS), period of invasive mechanical ventilation in days, medication need, hypoglycaemia, neonatal jaundice, sepsis and cardiovascular function.
Proportion of children with neurodevelopmental impairment | At two years of corrected age
  Neurodevelopmental impairment is defined as an abnormal test on Bayley III Dutch version (or version IV if available) (composite cognitive score < 85, composite motor score < 85), cerebral palsy, with a Gross Motor Function Classification System (GMFCS) grade > 1, hearing loss needing hearing aids, or severe visual loss (legally certifiable as blind or partially sighted) assessed at two years of corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Wessel Ganzevoort, MD PhD, Principal Investigator — Amsterdam UMC

IPD SHARING:
Plan to Share IPD: No
There is no current plan, but data will be available upon collaboration request